CLINICAL TRIAL: NCT00993785
Title: CoStar Catheter System Evaluation
Acronym: CONCISE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: CoStar Stent IDE failed to meet primary endpoint
Sponsor: Conor Medsystems (Industry)
Responsible Party: Sid Cohen, M.D., Cordis
Other Study IDs: CP-04
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Symptomatic Ischemic Heart Disease

ARMS (1):
- OTW Catheter System (Experimental)
  Interventions: Device: Costar Coronary Stent Delivery System

INTERVENTIONS:
Device: Costar Coronary Stent Delivery System

SUMMARY:
To evaluate product performance and safety of the Catheter Design for the treatment of a single coronary lesion.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years of age.
2. Eligible for percutaneous coronary intervention (PCI).
3. Documented stable or unstable angina pectoris (Canadian Cardiovascular Society Classification [CCS] 1, 2, 3, or 4), documented ischemia, or documented silent ischemia.
4. Left ventricular ejection fraction (LVEF) ≥25% documented within the last 6 weeks.
5. Acceptable candidate for coronary artery bypass graft surgery (CABG).
6. Patient understands the study requirements and the treatment procedures and provides written Informed Consent using a form that has been approved by the local Institutional Review Board or Ethics Committee before any study-specific tests or procedures are performed.
7. Willing to comply with all specified follow-up evaluations.

Inclusion Criteria (Angiographic):

1. A single de novo lesion per study subject may be treated with the study device.
2. Each target lesion may be composed of multiple lesions but must be completely coverable by one (1) study stent.
3. Cumulative target lesion length per vessel is ≤24 mm based on a visual estimate.
4. RVD of ≥2.5 mm to ≤3.0 mm based on a visual estimate.
5. Target lesion diameter stenosis ≥50% and <100% based on a visual estimate.
6. Target vessel has not undergone prior revascularization within the preceding 6 months.
7. Target lesion must be a minimum of 10 mm distance from any previously treated segment of the target vessel

Exclusion Criteria:

1. Known sensitivity to cobalt chromium, paclitaxel or polymeric matrices: PLGA.
2. Planned treatment with any other PCI device in the target vessel(s).
3. Acute MI within 72 hours prior to the index procedure as defined by the presence of a new pathologic Q wave, or creatinine kinase (CK) >2 times the laboratory upper limits of normal and elevated MB.
4. The patient is in cardiogenic shock.
5. Cerebrovascular Accident (CVA) within the past 6 months.
6. Acute or chronic renal dysfunction (creatinine >2.0 mg/dl or >150 µmol/L).
7. Contraindication to ASA or to clopidogrel.
8. Thrombocytopenia (platelet count <100, 000/mm3).
9. Active gastrointestinal (GI) bleeding within the past three months.
10. Any prior true anaphylactic reaction to contrast agents.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-02; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Herz-Kreislauf-Zentrum, Am Kurpark 1, Segeberger Kliniken GmbH, Germany